CLINICAL TRIAL: NCT04089605
Title: Ranibizumab and Dexamethasone Implant in Vitrectomized Eyes With Diabetic Macular Edema
Brief Title: Ranibizumab vs Dexamethasone Implant in Vitrectomized Eyes With Diabetic Macular Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jia-Kang Wang, Chief of the Vitreoretinal Section of Ophthalmology Department, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105136-E
Record Dates: First submitted 2019-09-01; First posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Macular Edema
Keywords: dexamethasone implant; vitrectomized; diabetic macular edema; ranibizumab
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; Ranibizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intravitreal dexamethasone implant (Experimental): The eyes undergo dexamethasone intravitreal implant 0.7 mg injections at baseline and every 3 or 4 months thereafter. Dexamethasone implants are re-injected in minimal 3-month interval if macular edema persisted or recurred with CFT more than 350 μm or manifestation of apparent submacular fluid and/or intramacular cysts. If DME subside with CFT less than 350 μm without accompanying fluid and cysts, repeated injection is mandatory in maximal 4-month interval.
  Interventions: Drug: dexamethasone implant
- intravitreal ranibizumab (Active Comparator): As for intravitreal ranibizumab 0.5 mg (IVR), we use OCT-guided treat-and-extend protocol for DME treatment after modifying the settings of TREX-DME study.4 The regimen include 3 monthly loading doses then extending the treatment injection interval one month more if CFT less than 350 μm without obvious submacular fluid and intramacular cysts. The injection interval shorten one month if CFT more than 350 μm or presence of obvious fluid and/or cysts. The patients are intentionally injected at most every 3 months even DME not existing.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: dexamethasone implant — intravitreal dexamethasone implant injections in vitrectomized patients with DME
  Other Names: Dexamethasone implants (Ozurdex®, Allergan Inc., Irvine, CA, USA)
  Arms: intravitreal dexamethasone implant
Drug: Ranibizumab — intravitreal ranibizumab injections in vitrectomized patients with DME
  Other Names: (Lucentis®, Ranibizumab (Novartis Pharma AG, Basel, Switzerland, and Genentech Inc., South San Francisco, CA, USA)
  Arms: intravitreal ranibizumab

SUMMARY:
Vitrectomy is required for removal of vitreous hemorrhage or retinal traction tissue in some patients with proliferative diabetic retinopathy. Post-vitrectomy macular edema may occur in these diabetic patients. Intravitreal injections of anti-VEGF agents or corticosteroid are required for treating diabetic macular edema (DME) in vitrectomized eyes. Intraocular levels of various cytokines may alter in the diabetic eyes following vitrectomy. Pharmacokinetics may be different between various intraocular agents in vitrectomized eyes. Herein our study will prospectively randomize to compare the clinical behavior between intravitreal ranibizumab (IVR) and intravitreal dexamethasone implant (IDI) in vitrectomized patients with DME. To our knowledge, it is the first study involving such subject.

DETAILED DESCRIPTION:
Vitrectomy is required for removal of vitreous hemorrhage or retinal traction tissue in some patients with proliferative diabetic retinopathy. Post-vitrectomy macular edema may occur in these diabetic patients. Intravitreal injections of anti-VEGF agents or corticosteroid are required for treating diabetic macular edema (DME) in vitrectomized eyes. Intraocular levels of various cytokines may alter in the diabetic eyes following vitrectomy. Pharmacokinetics may be different between various intraocular agents in vitrectomized eyes. Herein our study will prospectively randomize to compare the clinical behavior between intravitreal ranibizumab (IVR) and intravitreal dexamethasone implant (IDI) in vitrectomized patients with DME. To our knowledge, it is the first study involving such subject.

Pseudophakic vitrectomized eyes with treatment-naïve center-involved DME will be enrolled with one eye in each patient. They are randomized into one group receiving IDI every 3 to 4 months, and the other group undergoing IVR using 3 monthly plus treat-and-extend injections all with monthly follow-up for 6 months. Switch of intravitreal drugs or deferred macular laser is not allowed. Primary outcome measures include change in central foveal thickness (CFT) in 1 mm by spectral-domain optic coherence tomography, and best corrected visual acuity (BCVA) at Month 6. Primary outcome measures include change in CFT and BCVA at Month 6. Injection number, BCVA, CFT, post-injection complications, and IOP are recorded and compared with Wilcoxon signed rank test within the group and Wilcoxon rank sum test between groups. Fisher's exact test is used for categorical comparison between groups. P value less than 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* Glycosylated hemoglobin (HbA1c) less than 10.0%
* Best-corrected visual acuity (BCVA) between 20/400 to 20/40
* Central foveal thickness (CFT) more than 300 μm in the 1-mm central macular subfield on spectral domain optical coherence tomography (SD-OCT, CIRRUS™ HD-OCT 5000, Carl Zeiss Meditec Inc., Dublin, CA, USA) using 6 radial line scans through the fovea
* Macular leakage on fundus fluorescein angiography (HRA2, Heidelberg Engineering GmbH, Germany)
* The DME pattern can include submacular fluid, cystoid change, and diffuse macular thickening
* All have proliferative diabetic retinopathy treated by panretinal photocoagulation receiving prior vitrectomy without silicone oil or gas inside the vitreous cavity
* Prior intraocular surgery performed as least 3 months ago

Exclusion Criteria:

* Pregnant or nursing women
* The patients with the history of thromboembolic events or major surgery within the previous 3 months
* Presence of anterior chamber intraocular lens or subluxated/dislocated posterior chamber intraocular lens
* Presence of uncontrolled hypertension
* Known coagulation abnormalities or current use of anticoagulative medication other than aspirin
* Prior macular photocoagulation or photodynamic therapy
* Presence of active infectious disease or intraocular inflammation
* Intraocular pressure more than 20 mmHg or glaucoma history
* Presence of iris neovascularization/vitreous hemorrhage.
* The DME pattern with accompanying macular traction by epiretinal membrane or posterior hyaloid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
BCVA at Month 6 | Month 6
  best-corrected visual acuity (BCVA) at the end of intervention
CFT at Month 6 | Month 6
  central foveal thickness (CFT) at the end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Wen Chang, Ph. D., Study Chair — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang JK, Huang TL, Su PY, Chang PY. An updated review of long-term outcomes from randomized controlled trials in approved pharmaceuticals for diabetic macular edema. Eye Sci. 2015 Dec;30(4):176-83. PMID 27215008
- [Result] Sonoda S, Sakamoto T, Shirasawa M, Yamashita T, Otsuka H, Terasaki H. Correlation between reflectivity of subretinal fluid in OCT images and concentration of intravitreal VEGF in eyes with diabetic macular edema. Invest Ophthalmol Vis Sci. 2013 Aug 9;54(8):5367-74. doi: 10.1167/iovs.13-12382. PMID 23860753
- [Result] Muether PS, Droege KM, Fauser S. Vascular endothelial growth factor suppression times in patients with diabetic macular oedema treated with ranibizumab. Br J Ophthalmol. 2014 Feb;98(2):179-81. doi: 10.1136/bjophthalmol-2013-303954. Epub 2013 Nov 13. PMID 24227804